CLINICAL TRIAL: NCT00843700
Title: Effectiveness of IPT Adapted for Depressed Women With Trauma Histories in a Community Mental Health Center
Brief Title: Women's Depression Treatment Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nancy Talbot, Associate Professor, Department of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00020535; 1R01MH076928 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpersonal Psychotherapy (Experimental): Interpersonal Psychotherapy, 16 individual sessions within 32 weeks
  Interventions: Behavioral: Interpersonal Psychotherapy-Trauma in Community Settings
- Individual Psychotherapy (Active Comparator): Individual Psychotherapy, 16 individual sessions within 32 weeks
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy-Trauma in Community Settings — Interpersonal Psychotherapy-Trauma in Community Settings (IPT-TCS) is Interpersonal Psychotherapy with modifications specifically designed for the treatment of depressed patients with trauma histories seen in community settings.
  Arms: Interpersonal Psychotherapy
Behavioral: Treatment as Usual — Individual psychotherapy following usual care practice in a community mental health center.
  Arms: Individual Psychotherapy

SUMMARY:
The aim of the Women's Depression Treatment Study, based in a community mental health center, is to evaluate the effectiveness of Interpersonal Psychotherapy-Trauma in Community Settings (IPT-TCS) on improving depression and other psychological and social functioning. IPT-TCS is Interpersonal Psychotherapy with modifications specifically designed for the treatment of depressed patients with trauma histories seen in community settings.

DETAILED DESCRIPTION:
Evidence-based treatments for depression have rarely been studied in community settings where low-income and ethnic minority patients receive care. Among the most in need of effective treatments are depressed women with histories of early interpersonal trauma, who suffer disproportionate burden characterized by chronic depression, multiple comorbidities, and marked interpersonal difficulties. The aim of this randomized controlled trial (RCT), based in a community mental health center, is to evaluate the effectiveness of Interpersonal Psychotherapy-Trauma in Community Settings (IPT-TCS). IPT-TCS is Interpersonal Psychotherapy with modifications specifically designed for the treatment of depressed patients with trauma histories seen in community settings. This trial (n=180) will compare IPT-TCS to active treatment as usual (TAU) for women with major depression and histories of childhood sexual abuse. We hypothesize that IPT-TCS will be more effective than TAU in reducing depression at 32-weeks after treatment assignment. Improvements in social functioning, health-related functioning, post-traumatic stress symptoms, and mental health functioning are also expected. To monitor post-treatment course, outcome variables will be assessed at 6-month intervals over a 2-year period, and longer-term effects will be examined via repeated-measure analyses. This trial is designed to provide definitive results regarding the effectiveness of IPT-TCS compared to usual care in a community mental health center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current Major Depression
* History of sexual abuse prior to age 18

Exclusion Criteria:

* Bipolar disorder
* Psychosis or schizophrenia
* Active alcohol or substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM-IV diagnoses: Current Major Depression Module | 20 months

SECONDARY OUTCOMES:
Beck Depression Inventory | 20 months
Hamilton Rating Scale for Depression | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Talbot, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Talbot NL, Gamble SA. IPT for women with trauma histories in community mental health care. Journal of Contemporary Psychotherapy 38(1): 35-44, 2008.
- [Result] Lestrade KN, Talbot NL, Ward EA, Cort NA. High-risk sexual behaviors among depressed Black women with histories of intrafamilial and extrafamilial childhood sexual abuse. Child Abuse Negl. 2013 Jun;37(6):400-3. doi: 10.1016/j.chiabu.2013.01.007. Epub 2013 Mar 14. PMID 23499057
- [Derived] Glanton Holzhauer C, Duberstein P, Ward E, Talbot N. Reducing posttraumatic stress disorder symptom severity among depressed women with childhood sexual abuse histories in interpersonal psychotherapy-trauma: The role of improved social functioning. Psychol Trauma. 2024 Apr;16(Suppl 1):S285-S292. doi: 10.1037/tra0001293. Epub 2022 Jun 2. PMID 35653744
- [Derived] Cankaya B, Talbot NL, Ward EA, Duberstein PR. Parental sexual abuse and suicidal behaviour among women with major depressive disorder. Can J Psychiatry. 2012 Jan;57(1):45-51. doi: 10.1177/070674371205700108. PMID 22296967